CLINICAL TRIAL: NCT05534867
Title: Effects of Mandala Coloring on Anxiety in Pregnant Women: Randomized Controlled Experimental Study
Brief Title: Effects of Mandala Coloring on Anxiety in Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırklareli University (Other)
Collaborators: Cukurova University (Other)
Responsible Party: Principal Investigator, Ayca Solt Kirca, Asssistant professor, Kırklareli University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KırklareliAS-6
Record Dates: First submitted 2022-09-05; First posted 2022-09-10 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Anxiety; Pregnancy Related
Keywords: pregnancy; anxiety; mandala coloring
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mandala coloring group (Experimental): Mandala painting will be applied to pregnant women who have anxiety related to pregnancy.
  Interventions: Other: Mandala coloring
- Control group (No Intervention): Participants in this group will consist of people who do not routinely do any practice on their own to reduce anxiety symptoms.

INTERVENTIONS:
Other: Mandala coloring — Participants will be asked to choose the pages they want from 12 colored felt-tip pen paint sets and 16 mandala coloring pages given to each participant by the researcher for 1 month, 2 days a week, at any time of the day and for an average of 20-30 minutes each time, and paint them in the colors they want.
  Arms: Mandala coloring group

SUMMARY:
This research was planned as a randomized controlled experimental study in order to reduce the anxiety felt by expectant mothers in relation to pregnancy during pregnancy.

DETAILED DESCRIPTION:
Pregnancy is an important period in a woman's life in which she experiences different spiritual, physical and emotional experiences. While experiencing this process, women may face many factors that may affect their mental health, such as stress, anxiety and depression. When the literature is examined, it is stated that approximately 10% to 24.2% of pregnant women experience anxiety or stress during their pregnancy.It is very important to diagnose it in the early stages of pregnancy, as anxiety in pregnancy can have negative effects on maternal and newborn health, especially in the birth and postpartum period.

A number of alternatives have been found to reduce anxiety, one of which is using it in the form of art therapy.In the opinion of art psychotherapists, mandala painting is one of the main tools of other art psychotherapy techniques that focus on healing.A number of studies have been conducted to determine the effect of drawing or coloring a mandala on anxiety.

Amelia et al conducted research that proved that drawing and coloring mandalas effectively reduces students' anxiety levels. In Turkey, a study was conducted by Sezen and Ünsalver on the fear of childbirth in pregnant women, including art therapy. In the study, 7 types of art therapy were applied to the women, including listening to music and singing, making masks, drawing, making mandalas, making dolls, taking photographs and making collages. As a result of the research, it was determined that art therapy was effective in reducing anxiety.

When the studies are examined, there are studies on the application of mandala to reduce the anxiety felt by children in cancer patients, but there are no studies on reducing pregnancy-related anxiety of women during pregnancy. This research was planned as a randomized controlled experimental study in order to reduce the anxiety felt by expectant mothers in relation to pregnancy during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Ability to read and understand Turkish
* Being between the ages of 20-35,
* Single pregnancy
* Don't be primiparous
* Having 40 or more from STAI
* Volunteering to participate in the research
* Fully answering survey and scale forms.
* Being in the first, 2nd or 3rd trimester

Exclusion Criteria:

* Having been diagnosed with a risky pregnancy
* Unwilling to continue working
* Having a chronic disease (Diabetes, Hypertension, Thyroid etc.),
* Having any problem that prevents communication (such as hearing, speaking, and understanding abilities),
* Using one of the pharmacological or non-pharmacological methods to reduce anxiety and receiving psychiatric treatment (Pharmacotherapy or psychotherapy).
* Lack of a smart phone and internet

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 77 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Introductory Information form | between one to six months
  A form that includes questions about women's socio-demographic and pregnancy and characteristics.
the Spielberger State-Trait Anxiety Inventory (STAI) scale | between one to six months
  This scale, developed by Spielberg in 1973, consists of 20 questions. It is a 4-point Likert type scale (1=not at all, 4=very much). The lowest score that can be obtained from the scale is 20, and the highest score is 80. The higher the score is, the higher the anxiety level is. The alpha value of the scale is 0.86-.92.33. The validity and reliability study in our country was conducted by Oner et al., in 1983 and the alpha value was found between. The scale that will be used to evaluate the state and trait anxiety of pregnant women. As the score increases, it is determined that the anxiety is higher.
Pregnancy-related anxiety scale | between one to six months
  This scale was developed by Brunton, whose validity and reliability in Turkish were made by Şolt and Gül. As the score obtained from the scale increases, the level of pregnancy-related anxiety increases. It will be used to assess pregnancy-related anxiety. As the score obtained in the scale consisting of 9 sub-dimensions increases, it is determined that the anxiety of the pregnant woman is also higher.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Dağlı, Phd, Principal Investigator — Cukurova University; AYÇA ŞOLT KIRCA, Phd, Study Director — Kırklareli University
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Solt Kirca A, Dagli E. The effect of mandala coloring on pregnancy-related anxiety. Eur J Obstet Gynecol Reprod Biol. 2024 Jan;292:251-258. doi: 10.1016/j.ejogrb.2023.11.035. Epub 2023 Dec 1. PMID 38056411